CLINICAL TRIAL: NCT01174342
Title: The Effect of Child Delivery on the Intraocular Pressure
Brief Title: Effect of Child Delivery on Intraocular Pressure
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 099-2010mmc
Record Dates: First submitted 2010-08-01; First posted 2010-08-03 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Intraocular Pressure; Delivery, Obstetric
Keywords: Intraocular pressure; Ocular tonometry; Obstetric delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Healthy pregnant women

SUMMARY:
The purpose of this study is to evaluate the effect of child delivery on the intraocular pressure in healthy women.

DETAILED DESCRIPTION:
Little is known about the changes in intraocular pressure (IOP) during child delivery. During labor there are several stages which are accompanied by many physiological changes and pharmacological interventions that may potentially influence the IOP. Among these are delivery position (lying versus sitting or kneeling), vascular changes and pharmacological effects (anesthetic agents, oxytocin and other drugs). The purpose of this study is to evaluate the effect of child delivery on the intraocular pressure (IOP) in healthy women. This will expend our understanding of the physiology of labor and its effect on the eye and it may serve as basis to determine the management of labor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Pregnant women admitted to the labor room.
* Healthy women that do not take any systemic medications.
* No known ocular condition, except for refraction errors, strabismus or amblyopia.
* Eligible women who are able to sign an informed consent form.

Exclusion Criteria:

* Family history of glaucoma (first degree relatives).
* Known allergic reaction to local anesthesia (oxybuprocaine hydrochloride).
* Women who are unable to sign an informed consent form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy women candidate for chlid delivery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fani Segev, M.D., Study Chair — Meir Medical Center; Noa Geffen, M.D., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy pregnant women candidates for vaginal delivery were recruited at their acceptance to the delivery room, between August 2010 and August 2012, in a single center (Meir medical center).
Pre-assignment Details: No relevant pre-assignment details exist.
Groups:
- Healthy Pregnant Women: Healthy pregnant women candidates for vaginal delivery.
Period: Overall Study
Arm/Group | Healthy Pregnant Women
Started | 30
Completed | 26
Not Completed | 4
Not completed — Conversion to cesarean section | 4

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Pregnant Women
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  Israel | 30

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Intraocular pressure during different stages of child delivery.
Time Frame: During child delivery
Population: We included in the analysis all women completing vaginal delivery that had measurements of their intraocular pressure during most stages of labor.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Healthy Pregnant Women
Number analyzed (Participants) | 26
mm Hg
  Intraocular pressure on admission | 11.8 (3.6)
  Intraocular pressure in Stage 1 latent phase | 11.9 (3.3)
  Intraocular pressure in Stage 1 active phase | 11.8 (2.9)
  Intraocular pressure in Stage 2 | 12.1 (3.1)
  Intraocular pressure in Stage 3 | 12.2 (4)
  Intraocular pressure 24 hours postpartum | 11.9 (2.4)
  Intraocular pressure 48 hours postpartum | 13.2 (2.3)

ADVERSE EVENTS:
Arm/Group | Healthy Pregnant Women
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
The number of participants was small due to difficulties in recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes